CLINICAL TRIAL: NCT02686658
Title: A Phase 2/3 Randomized, Double-Masked, Controlled Trial to Assess the Safety and Efficacy of Intravitreous Administration of Zimura™ (Anti-C5 Aptamer) in Patients With Geographic Atrophy Secondary to Dry Age-Related Macular Degeneration
Brief Title: Zimura in Participants With Geographic Atrophy Secondary to Dry Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IVERIC bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPH2003; 2015-003991-56 (EudraCT Number)
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Geographic Atrophy; Dry Age-Related Macular Degeneration
Keywords: Geographic Atrophy (GA); Dry age-related macular degeneration; AMD; Zimura (previous name); Anti-inflammatory; complement factor C5 inhibitor; ARC1905; avacincaptad pegol
MeSH Terms: conditions — Geographic Atrophy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Reading Center team and Sponsor were also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Avacincaptad Pegol 1 mg [Part 1] (Experimental): Participants received 1 mg of Avacincaptad Pegol in the study eye administered via IVT injection (50 µL) on Day 1 and monthly up to 18 months.
  Interventions: Drug: Avacincaptad Pegol
- Avacincaptad Pegol 2 mg [Part 1] (Experimental): Participants received 2 mg of Avacincaptad Pegol in the study eye administered via IVT injection (100 µL) on Day 1 and monthly up to 18 months.
  Interventions: Drug: Avacincaptad Pegol
- Sham [Part 1] (Sham Comparator): Participants received a Sham injection of an empty, needleless syringe administered in the study eye on Day 1 and monthly up to 18 months.
  Interventions: Other: Sham
- Avacincaptad Pegol 2 mg (Avacincaptad Pegol 2mg+Sham) [Part 2] (Experimental): Participants received 2 mg of Avacincaptad Pegol in the study eye administered via IVT injection (100 µL) and a subsequent Sham administration on Day 1 and monthly up to 18 months.
  Interventions: Drug: Avacincaptad Pegol; Other: Sham
- Avacincaptad Pegol 4 mg (Avacincaptad Pegol 2mg+Avacincaptad Pegol 2mg) [Part 2] (Experimental): Participants received 4 mg of Avacincaptad Pegol in the study eye administered via two consecutive IVT injections (2 x 100 µL) on Day 1 and monthly up to 18 months.
  Interventions: Drug: Avacincaptad Pegol
- Sham (Sham+Sham) [Part 2] (Sham Comparator): Participants received two consecutive Sham injections of empty, needleless syringes administered in the study eye on Day 1 and monthly up to 18 months.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Avacincaptad Pegol — Avacincaptad Pegol 20 mg/mL solution for intravitreal (IVT) injection
  Other Names: Zimura (previous name); IZERVAY; ARC1905
  Arms: Avacincaptad Pegol 1 mg [Part 1]; Avacincaptad Pegol 2 mg (Avacincaptad Pegol 2mg+Sham) [Part 2]; Avacincaptad Pegol 2 mg [Part 1]; Avacincaptad Pegol 4 mg (Avacincaptad Pegol 2mg+Avacincaptad Pegol 2mg) [Part 2]
Other: Sham — The Sham procedure included the blunt opening of an empty, needleless syringe barrel placed on the conjunctiva in the inferotemporal quadrant of the eyeball to simulate the pressure of an injection.
  Arms: Avacincaptad Pegol 2 mg (Avacincaptad Pegol 2mg+Sham) [Part 2]; Sham (Sham+Sham) [Part 2]; Sham [Part 1]

SUMMARY:
The objectives of this study were to evaluate the safety and efficacy of Zimura intravitreal (IVT) administration when administered in participants with geographic atrophy (GA) secondary to dry age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Participants will receive monthly intravitreal injections of Zimura or Sham for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants of either gender aged ≥ 50 years
* Diagnosis of Non-foveal GA secondary to dry AMD

Exclusion Criteria:

* Evidence of Choroidal Neovascularization (CNV)
* GA secondary to any condition other than AMD
* Any prior treatment for AMD or any prior intravitreal treatment for any indication in either eye, except oral supplements of vitamins and minerals
* Any intraocular surgery or thermal laser within three (3) months of trial entry
* Any prior thermal laser in the macular region, regardless of indication
* Any ocular or periocular infection in the twelve (12) weeks
* Previous therapeutic radiation in the region of the study eye
* Any sign of diabetic retinopathy in either eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (51):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Campbell, California
  - Fresno, California
  - Fullerton, California
  - La Jolla, California
  - Mountain View, California
  - Redlands, California
  - Sacramento, California
  - Santa Ana, California
  - Denver, Colorado
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Melbourne, Florida
  - St. Petersburg, Florida
  - Stuart, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - West Des Moines, Iowa
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Grand Rapids, Michigan
  - Henderson, Nevada
  - Reno, Nevada
  - Rochester, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - West Mifflin, Pennsylvania
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Abilene, Texas
  - Amarillo, Texas
  - Austin, Texas
  - Grapevine, Texas
  - Houston, Texas
  - The Woodlands, Texas
  - Willow Park, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
- Clinical hospital center Osijek, Osijek, Croatia
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno
  - Faculty Hospital Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Axon Clinical SRO, Prague
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Dr.Kai Noor Eye Clinic, Tallinn
- Hungary (6):
  - Peterfy Korhaz-Rendelointezet Orszagos Traumatologiai Intezet, Budapest
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
  - Veszprém
- Israel (6):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Result] Jaffe GJ, Westby K, Csaky KG, Mones J, Pearlman JA, Patel SS, Joondeph BC, Randolph J, Masonson H, Rezaei KA. C5 Inhibitor Avacincaptad Pegol for Geographic Atrophy Due to Age-Related Macular Degeneration: A Randomized Pivotal Phase 2/3 Trial. Ophthalmology. 2021 Apr;128(4):576-586. doi: 10.1016/j.ophtha.2020.08.027. Epub 2020 Sep 1. PMID 32882310
- [Derived] Corradetti G, Karamat A, Srinivas S, Lindenberg S, Velaga SB, Corvi F, Attiku Y, Nittala MG, Desai D, Zhu L, Abulon D, Sadda SR. Progression to complete retinal pigment epithelium and outer retinal atrophy (cRORA): post hoc analysis of the GATHER1 trial. Graefes Arch Clin Exp Ophthalmol. 2025 Mar;263(3):669-677. doi: 10.1007/s00417-024-06676-7. Epub 2024 Nov 14. PMID 39538001
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26398&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study participants are planned to receive 18 monthly intravitreal injections of Zimura and/or Sham in a single designated study eye. The study eye is designated by the Investigator prior to first administration of study drug and does not change throughout the duration of study participation.
Groups:
- Zimura 1 mg [Part 1]: Participants received 1 mg of Zimura in the study eye administered via intravitreal (IVT) injection on Day 1 and monthly up to 18 months.
- Zimura 2 mg [Part 1]: Participants received 2 mg of Zimura in the study eye administered via IVT injection on Day 1 and monthly up to 18 months.
- Zimura 2 mg (Zimura 2mg+Sham) [Part 2]: Participants received 2 mg of Zimura in the study eye administered via IVT injection and a Sham administration on Day 1 and monthly up to 18 months.
- Zimura 4 mg (Zimura 2mg+Zimura 2mg) [Part 2]: Participants received 4 mg of Zimura in the study eye administered via 2 IVT injections on Day 1 and monthly up to 18 months.
- Sham (Sham+Sham) [Part 2]: Participants received 2 Sham injections of empty, needleless syringes administered in the study eye on Day 1 and monthly up to 18 months.
Period: Overall Study
Arm/Group | Zimura 1 mg [Part 1] | Zimura 2 mg [Part 1] | Sham [Part 1] | Zimura 2 mg (Zimura 2mg+Sham) [Part 2] | Zimura 4 mg (Zimura 2mg+Zimura 2mg) [Part 2] | Sham (Sham+Sham) [Part 2]
Started | 26 | 25 | 26 | 42 | 83 | 84
Month 12 | 23 | 19 | 19 | 34 | 56 | 72
Completed | 22 | 18 | 17 | 30 | 46 | 68
Not Completed | 4 | 7 | 9 | 12 | 37 | 16
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Investigator decision | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Sponsor decision | 1 | 2 | 1 | 5 | 13 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 5 | 4 | 4 | 17 | 8
Not completed — Placed in hospice care | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant non-compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Concern over coronavirus disease care | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zimura 1 mg [Part 1] | Zimura 2 mg [Part 1] | Sham [Part 1] | Zimura 2 mg (Zimura 2mg+Sham) [Part 2] | Zimura 4 mg (Zimura 2mg+Zimura 2mg) [Part 2] | Sham (Sham+Sham) [Part 2] | Total
Number analyzed (Participants) | 26 | 25 | 26 | 42 | 83 | 84 | 286
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 2 | 6 | 5 | 4 | 24
  >=65 years | 23 | 21 | 24 | 36 | 78 | 80 | 262
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 18 | 27 | 58 | 61 | 197
  Male | 11 | 7 | 8 | 15 | 25 | 23 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 25 | 24 | 25 | 42 | 82 | 83 | 281
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 25 | 25 | 25 | 42 | 82 | 82 | 281
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geographic Atrophy as Measured by Fundus Autofluorescence
Description: The least squares mean change in geographic atrophy (GA) from baseline to Month 12 was measured by fundus autofluorescence (FAF). The square root of the GA area was used in the analysis. Per statistical analysis plan, only the Zimura 2 mg and 4 mg groups were evaluated for this primary endpoint; the Zimura 1 mg group was for descriptive purposes only.
Time Frame: Baseline and 12 months
Population: This study was conducted in 2 Parts. The analyses were based on comparisons of Zimura 2mg vs. Sham control and Zimura 4mg vs. Sham control. For comparison of Zimura 2mg vs. Sham control, participants randomized in Part 1 were combined with participants randomized in Part 2. Comparison of Zimura 4mg vs. Sham control was based on participants randomized in Part 2 only.
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Groups:
- Zimura 2 mg [Part 1 & Part 2 Combined]: Participants received 2 mg of Zimura in the study eye administered via IVT injection (or via IVT injection and a Sham administration) on Day 1 and monthly up to 18 months.
- Sham [Part 1 & Part 2 Combined]: Participants received a Sham injection (or 2 Sham injections) of an empty, needleless syringe administered in the study eye on Day 1 and monthly up to 18 months.
- Zimura 4 mg [Part 2]: Participants received 4 mg of Zimura in the study eye administered via 2 IVT injections on Day 1 and monthly up to 18 months.
- Sham [Part 2]: Participants received 2 Sham injections of empty, needleless syringes administered in the study eye on Day 1 and monthly up to 18 months.
Arm/Group | Zimura 2 mg [Part 1 & Part 2 Combined] | Sham [Part 1 & Part 2 Combined] | Zimura 4 mg [Part 2] | Sham [Part 2]
Number analyzed (Participants) | 67 | 110 | 83 | 84
millimeters (mm) | 0.292 (0.077) | 0.402 (0.075) | 0.321 (0.074) | 0.444 (0.072)
Statistical Analysis 1: Comparison: Zimura 2 mg [Part 1 & Part 2 Combined] vs Sham [Part 1 & Part 2 Combined]; Difference in least squares means between groups calculated as (Sham) minus (Zimura); Test type: Other — Model for repeated measures (MRM) and square root transformation was used to compare the treatment groups; p = 0.0072, Model for repeated measures (MRM); Least Squares Mean Difference = 0.110
Statistical Analysis 2: Comparison: Zimura 4 mg [Part 2] vs Sham [Part 2]; Difference in least squares means between groups calculated as (Sham) minus (Zimura); Test type: Other — Model for repeated measures (MRM) and square root transformation was used to compare treatment groups; p = 0.0051, Model for repeated measures (MRM); Least Squares Mean Difference = 0.124

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity Using Early Treatment Diabetic Retinopathy Study Letters
Description: The least squares mean change in best-corrected visual acuity (BCVA) from baseline to Month 12 was measured using early treatment diabetic retinopathy study [ETDRS] letters. Per statistical analysis plan, only the Zimura 2 mg and 4 mg groups were evaluated for the secondary endpoints; the Zimura 1 mg group was for descriptive purposes only.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | Zimura 2 mg [Part 1 & Part 2 Combined] | Sham [Part 1 & Part 2 Combined] | Zimura 4 mg [Part 2] | Sham [Part 2]
Number analyzed (Participants) | 67 | 110 | 83 | 84
ETDRS Letters | -7.90 (2.66) | -9.29 (2.59) | -3.79 (3.11) | -3.51 (2.99)
Statistical Analysis 1: Comparison: Zimura 2 mg [Part 1 & Part 2 Combined] vs Sham [Part 1 & Part 2 Combined]; Difference in least squares mean between groups calculated as (Zimura) minus (Sham); Test type: Other — Model for repeated measures (MRM) was used to compare the treatment groups; p = 0.3464, Model for repeated measures (MRM); Least Squares Mean Difference = 1.39
Statistical Analysis 2: Comparison: Zimura 4 mg [Part 2] vs Sham [Part 2]; Difference in least squares mean between groups calculated as (Zimura) minus (Sham); Test type: Other — Model for repeated measures (MRM) was used to compare the treatment groups; p = 0.8830, Model for repeated measures (MRM); Least Squares Mean Difference = -0.28

3. Secondary Outcome: Change From Baseline in Low Luminance BCVA Using Early Treatment Diabetic Retinopathy Study Letters
Description: The least squares mean change in low luminance (LL) BCVA from baseline to Month 12 was measured using ETDRS letters. Per statistical analysis plan, only the Zimura 2 mg and 4 mg groups were evaluated for the secondary endpoints; the Zimura 1 mg group was for descriptive purposes only.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | Zimura 2 mg [Part 1 & Part 2 Combined] | Sham [Part 1 & Part 2 Combined] | Zimura 4 mg [Part 2] | Sham [Part 2]
Number analyzed (Participants) | 67 | 110 | 83 | 84
ETDRS Letters | -1.03 (3.40) | -1.41 (3.30) | 1.53 (3.53) | 2.97 (3.39)
Statistical Analysis 1: Comparison: Zimura 2 mg [Part 1 & Part 2 Combined] vs Sham [Part 1 & Part 2 Combined]; Difference in least squares mean between groups calculated as (Zimura) minus (Sham); Test type: Other — Model for repeated measures (MRM) was used to compare the treatment groups; p = 0.8405, Model for repeated measures (MRM); Least Squares Mean Difference = 0.38
Statistical Analysis 2: Comparison: Zimura 4 mg [Part 2] vs Sham [Part 2]; Difference in least squares mean between groups calculated as (Zimura) minus (Sham); Test type: Other — Model for repeated measures (MRM) was used to compare the treatment groups; p = 0.5017, Model for repeated measures (MRM); Least Squares Mean Difference = -1.44

ADVERSE EVENTS:
Time Frame: Adverse events were recorded starting at Day 1 after the first dose of study drug and continuing until 30 days after the last dose or until the last follow-up visit required by the protocol, whichever comes later (up to approximately 18 months from first dose).
Description: The analysis population for all-cause mortality, serious adverse events (SAEs), and non-serious adverse events (NSAEs) consisted of all participants who received at least one dose of study treatment. Participants who received an injection of Zimura during this study were analyzed in the appropriate Zimura group according to the actual injections received.
Groups:
- Zimura (Any Dose) [Part 1 & Part 2 Combined]: Participants received a 1 mg, 2 mg, or 4 mg dose of Zimura in the study eye administered via 1 or 2 IVT injection(s) (or via IVT injection and a Sham administration) on Day 1 and monthly up to 18 months.
- Sham [Part 1 & Part 2 Combined]: Participants received a Sham injection (or 2 Sham injections) of empty, needleless syringes administered in the study eye on Day 1 and monthly up to 18 months.
Arm/Group | Zimura 1 mg [Part 1] | Zimura 2 mg [Part 1] | Sham [Part 1] | Zimura 2 mg (Zimura 2mg+Sham) [Part 2] | Zimura 4 mg (Zimura 2mg+Zimura 2mg) [Part 2] | Sham (Sham+Sham) [Part 2] | Zimura (Any Dose) [Part 1 & Part 2 Combined] | Sham [Part 1 & Part 2 Combined]
All-Cause Mortality (participants affected / at risk) | 1/26 | 0/25 | 0/26 | 1/42 | 1/83 | 1/84 | 3/176 | 1/110
Serious Adverse Events (participants affected / at risk) | 3/26 | 4/25 | 7/26 | 8/42 | 21/83 | 21/84 | 36/176 | 28/110
Other Adverse Events (participants affected / at risk) | 13/26 | 13/25 | 10/26 | 34/42 | 66/83 | 49/84 | 126/176 | 59/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zimura 1 mg [Part 1] (N=26) | Zimura 2 mg [Part 1] (N=25) | Sham [Part 1] (N=26) | Zimura 2 mg (Zimura 2mg+Sham) [Part 2] (N=42) | Zimura 4 mg (Zimura 2mg+Zimura 2mg) [Part 2] (N=83) | Sham (Sham+Sham) [Part 2] (N=84) | Zimura (Any Dose) [Part 1 & Part 2 Combined] (N=176) | Sham [Part 1 & Part 2 Combined] (N=110)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Optic ischaemic neuropathy* (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 — * included study and fellow eye events
Retinal detachment* (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 — * included study and fellow eye events
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 1 | 4 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zimura 1 mg [Part 1] (N=26) | Zimura 2 mg [Part 1] (N=25) | Sham [Part 1] (N=26) | Zimura 2 mg (Zimura 2mg+Sham) [Part 2] (N=42) | Zimura 4 mg (Zimura 2mg+Zimura 2mg) [Part 2] (N=83) | Sham (Sham+Sham) [Part 2] (N=84) | Zimura (Any Dose) [Part 1 & Part 2 Combined] (N=176) | Sham [Part 1 & Part 2 Combined] (N=110)
Conjunctival haemorrhage * (Eye disorders) | 2 | 2 | 1 | 9 | 28 | 12 | 41 | 13 — * included study and fellow eye events
Neovascular age-related macular degeneration* (Eye disorders) | 3 | 2 | 2 | 7 | 11 | 2 | 23 | 4 — * included study and fellow eye events
Conjunctival hyperaemia* (Eye disorders) | 0 | 0 | 0 | 3 | 9 | 4 | 12 | 4 — * included study and fellow eye events
Punctate keratitis* (Eye disorders) | 0 | 0 | 0 | 4 | 6 | 8 | 10 | 8 — * included study and fellow eye events
Eye pain* (Eye disorders) | 0 | 1 | 0 | 1 | 8 | 3 | 10 | 3 — * included study and fellow eye events
Vitreous detachment* (Eye disorders) | 3 | 0 | 0 | 2 | 4 | 6 | 9 | 6 — * included study and fellow eye events
Cataract* (Eye disorders) | 2 | 0 | 1 | 4 | 2 | 5 | 8 | 6 — * included study and fellow eye events
Visual acuity reduced* (Eye disorders) | 0 | 2 | 0 | 2 | 3 | 8 | 7 | 8 — * included study and fellow eye events
Conjunctival oedema* (Eye disorders) | 0 | 0 | 0 | 2 | 5 | 4 | 7 | 4 — * included study and fellow eye events
Choroidal neovascularization* (Eye disorders) | 1 | 0 | 0 | 0 | 5 | 3 | 6 | 3 — * included study and fellow eye events
Eye irritation* (Eye disorders) | 0 | 0 | 1 | 3 | 2 | 4 | 5 | 5 — * included study and fellow eye events
Posterior capsule opacification* (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2 — * included study and fellow eye events
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 7 | 10 | 8 | 19 | 10
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 4 | 3 | 5 | 11 | 5
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 2 | 3 | 3 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 5 | 2 | 8 | 2
Influenza (Infections and infestations) | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 2 | 3 | 2
Intraocular pressure increased (Investigations) | 1 | 2 | 0 | 4 | 19 | 1 | 26 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 8 | 6 | 7 | 14 | 7
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 3 | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 2 | 0 | 3 | 2
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 3 | 2 | 4 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 2
Dementia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual site or investigator may publish or present any results from the trial until a joint, multi-center publication of the trial results is made by Sponsor in conjunction with various participating investigators and appropriate sites contributing data and comments. Subsequently, individual investigators may request to publish or present results from the trial; however approval will be at the sole discretion of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT02686658/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT02686658/SAP_001.pdf